CLINICAL TRIAL: NCT03090477
Title: Impact of a Pharmaceutical Care Model in the Management of Chronic Myeloid Leukemia Patients. A Randomised Control Trial
Brief Title: Impact of a Pharmaceutical Care Model in the Management of Chronic Myeloid Leukemia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSI University (Other)
Collaborators: University of Malaya (Other); Ampang Hospital, Malaysia (Unknown)
Responsible Party: Principal Investigator, Bee kim Tan, Lecturer, UCSI University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NMRR23315
Record Dates: First submitted 2017-03-18; First posted 2017-03-24 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Medication Adherence
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Medication Adherence | interventions — Pharmaceutical Services

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmaceutical care and adherence aids (Experimental)
  Interventions: Behavioral: Pharmaceutical care and adherence aids
- Control (dispensing of TKI & instruction about administration) (No Intervention)

INTERVENTIONS:
Behavioral: Pharmaceutical care and adherence aids — Medication review including drug-interaction check, individual patient counseling to improve understanding of treatment rationale and to elicit and address treatment-related concerns, provision of information booklets and adherence aids (calender blister packaging and smartphone medication reminder application), phone calls and face-to-face visits to follow-up on medication-related issues scheduled over a period of 6 months.
  Arms: Pharmaceutical care and adherence aids

SUMMARY:
Owing to effective treatment with tyrosine kinase inhibitors (TKIs), chronic myeloid leukemia (CML) has become a chronic disease with a rising prevalence globally. Although the possibility of stopping TKI therapy in CML patients who have achieved deep molecular responses is a topic of active debate and investigation, life-long treatment remains the current standard of care. It has been estimated that 3% to 56% of CML patients are not adherent to their prescribed TKI therapy. Poor adherence to TKIs could compromise the control of CML, and contributes to poorer survival. CML patients on long-term TKI therapy are prone to developing certain medication-related issues such as adverse reactions and drug interactions.Occurrence of adverse reactions even at low grades, has been shown to impact CML patient's health-related quality of life (HRQoL) and adherence to treatment. However, there is no prospective high quality evidence showing adherence to TKIs and the associated clinical outcomes can be improved in CML patients. Therefore, the investigators hypothesize that medication management intervention by pharmacist might improve adherence to TKIs, and translate into better disease response and HRQoL in CML patients, when compared to control arm who receive standard pharmacy service.

ELIGIBILITY:
Inclusion Criteria:

* has a confirmed diagnosis of Philadelphia chromosome positive CML
* has a detectable BCR-ABL1 mRNA
* has been taking TKI for at least 3 months
* able to speak and read English, Malay or Mandarin

Exclusion Criteria:

* with cognitive deficit or psychiatric disorders
* in advanced phase of CML where TKI is transitory to hematologic stem cell transplant
* history of hematologic stem cell transplant
* pregnant or plan to conceive in the next 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2018-06-24 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in percentage of patients who adhere to prescribed TKI therapy | Evaluated at 2 time frame, (a) Immediate effect of intervention: 1-3 months pre-intervention until 6 months after starting intervention; (b) long-term effect of intervention: 1-3 months pre-intervention until 6 months after the end of intervention
  Adherence is defined as having an medication possession ratio (MPR) of greater than 90% (calculated as days' supply of TKI dispensed divided by number of days of the study period) from electronic prescription refill database system

SECONDARY OUTCOMES:
Changes in percentage of patients who achieve major/deep molecular response to TKI | Evaluated at 2 time frame, (a) 0-3 months pre-intervention until 6 months after starting intervention; (b) 0-3 months pre-intervention until 6 months after the end of intervention
  Molecular response is determined as log-reduction of BCR-ABL1 mRNA by polymerase chain reaction (PCR) in international scale (IS)
Mean changes in health-related quality of life status | Evaluated at 2 time frame, (a) 1 week pre-intervention until 6 months after starting intervention; (b) 1 week pre-intervention until 6 months after the end of intervention
  HRQoL is determined as patient-reported score on EORTC QLQ-C30 and CML24 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bee Kim Tan, RPh, Principal Investigator — UCSI University
Locations (2):
- Malaysia (2):
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Ampang hospital, Ampang, Selangor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marin D, Bazeos A, Mahon FX, Eliasson L, Milojkovic D, Bua M, Apperley JF, Szydlo R, Desai R, Kozlowski K, Paliompeis C, Latham V, Foroni L, Molimard M, Reid A, Rezvani K, de Lavallade H, Guallar C, Goldman J, Khorashad JS. Adherence is the critical factor for achieving molecular responses in patients with chronic myeloid leukemia who achieve complete cytogenetic responses on imatinib. J Clin Oncol. 2010 May 10;28(14):2381-8. doi: 10.1200/JCO.2009.26.3087. Epub 2010 Apr 12. PMID 20385986
- [Background] Lam MS, Cheung N. Impact of oncology pharmacist-managed oral anticancer therapy in patients with chronic myelogenous leukemia. J Oncol Pharm Pract. 2016 Dec;22(6):741-748. doi: 10.1177/1078155215608523. Epub 2015 Sep 28. PMID 26419691
- [Background] Noens L, Hensen M, Kucmin-Bemelmans I, Lofgren C, Gilloteau I, Vrijens B. Measurement of adherence to BCR-ABL inhibitor therapy in chronic myeloid leukemia: current situation and future challenges. Haematologica. 2014 Mar;99(3):437-47. doi: 10.3324/haematol.2012.082511. PMID 24598855
- [Background] Moon JH, Sohn SK, Kim SN, Park SY, Yoon SS, Kim IH, Kim HJ, Kim YK, Min YH, Cheong JW, Kim JS, Jung CW, Kim DH. Patient counseling program to improve the compliance to imatinib in chronic myeloid leukemia patients. Med Oncol. 2012 Jun;29(2):1179-85. doi: 10.1007/s12032-011-9926-8. Epub 2011 Apr 7. PMID 21472487
- [Background] Kekale M, Peltoniemi M, Airaksinen M. Patient-reported adverse drug reactions and their influence on adherence and quality of life of chronic myeloid leukemia patients on per oral tyrosine kinase inhibitor treatment. Patient Prefer Adherence. 2015 Dec 8;9:1733-40. doi: 10.2147/PPA.S92125. eCollection 2015. PMID 26677317
- [Derived] Tan BK, Chua SS, Chen LC, Chang KM, Balashanker S, Bee PC. Efficacy of a medication management service in improving adherence to tyrosine kinase inhibitors and clinical outcomes of patients with chronic myeloid leukaemia: a randomised controlled trial. Support Care Cancer. 2020 Jul;28(7):3237-3247. doi: 10.1007/s00520-019-05133-0. Epub 2019 Nov 16. PMID 31734798